CLINICAL TRIAL: NCT02831114
Title: Evaluating the Effects of Acupuncture in the Treatment of Taxane Induces Peripheral Neuropathy (TIPN)
Brief Title: Evaluating the Effects of Acupuncture in the Treatment of Taxane Induces Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00038410
Record Dates: First submitted 2016-05-25; First posted 2016-07-13 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2016-05

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The nine participants in the intervention arm will receive 18 acupuncture treatments over the course of 12 weeks (2 treatments per week for 6 weeks and 1 treatment per week for 6 weeks). They will undergo assessments at baseline, 6 weeks, and 12 weeks through the use of questionnaires and blood tests. The participants will also be allowed to continue their conventional therapy for TIPN.
  Interventions: Other: Acupuncture
- Control (No Intervention): The nine participants in this arm will undergo the same assessments as the intervention arm at baseline, 6 weeks, and 12 weeks. They will not receive any acupuncture treatments during this time, but will be allowed to continue their conventional therapy. The control arm will be offered the same 18 acupuncture treatments after a wait of at least 12 weeks.

INTERVENTIONS:
Other: Acupuncture — Acupuncture uses tiny needles to promote blood flow, nervous system signaling, and brings the body back into homeostasis which the state of optimum functioning. Treatment for taxane induced peripheral neuropathy will consist of traditional acupuncture and will use points located in the foot (SP 3, ST 41, LR 3, K 3, GB 41), knee (SP 9, ST 36, K 10, GB 34), and arm (LI 11). Participants will continue to take their conventional therapy. Each acupuncture treatment will take place at Oriental Medicine Associates with trained acupuncturist, William Hendry. Each session should last about 30 minutes.
  Arms: Intervention

SUMMARY:
Taxane Induced Peripheral Neuropathy (TIPN) is a major dose limiting side effect of taxane chemotherapies and it often reduces the success of the patient treatment. Treating TIPN is difficult and at this time conventional treatment is primarily limited to the global use of antidepressants and anticonvulsants. Acupuncture treatment has been used for symptom improvement in patients with peripheral neuropathy caused by HIV and diabetes mellitus; however, few studies have evaluated acupuncture as a viable treatment for taxane induced peripheral neuropathy. This study will enroll female breast cancer survivors at the Greenville Health System Cancer Institute Center for Integrative Oncology and Survivorship to assess whether acupuncture holds any therapeutic benefit for TIPN and how it influences the mechanisms underlying resolution of TIPN. This would provide critical validation of acupuncture and increase potential for other forms of chemotherapy induced peripheral neuropathy.

DETAILED DESCRIPTION:
Taxane induced peripheral neuropathy (TIPN) affects many female breast cancer survivors treated with taxane chemotherapies. This condition can include symptoms ranging from minor loss of sensory function, numbness and mild paresthesia to frank pain including burning or tingling sensation or shooting neuropathic pain. Treating TIPN is difficult and at this time conventional treatment is primarily limited to the use of antidepressants and anticonvulsants, both of which have significant efficacy and safety issues with often little reduction in TIPN. The mechanisms of taxane induced peripheral tissue damage are becoming clearer allowing for the potential to develop specific interventions to resolve pain associated with this class of drug. Acupuncture treatment has been used for symptom improvement in patients with peripheral neuropathy caused by HIV and diabetes mellitus; however, few studies have evaluated acupuncture as a viable treatment for taxane induced peripheral neuropathy. Moreover, there has been little research considering the biological effect of acupuncture treatment related to the mechanisms of pain resolution. This study will enroll female breast cancer survivors at the Greenville Health System Cancer Institute Center for Integrative Oncology and Survivorship undergo an acupuncture protocol consisting of traditional acupuncture points used for neuropathic pain. This is a prospective, randomized, controlled trial that will consist of two arms. The two arms will consist of 1) acupuncture plus conventional therapy and 2) conventional therapy only (n= 9 participants in each arm). Arm 1 will receive a traditional manual acupuncture protocol twice a week for 6 weeks and once a week for 6 weeks in conjunction with standard of care treatment. Arm 2 will receive standard of care treatment only; acupuncture will be offered to these individuals after a 12 week waitlist. The 18 participants will start an individualized 12 week study schedule and will be recruited over a 4 month time period. This study will assess severity of pain, inflammatory biomarkers, and circulating levels of mitochondrial DNA at baseline, 6 weeks, and 12 weeks for both arms through questionnaires and blood tests. Results of the study will further clarify acupuncture's role as a therapeutic modality for managing pain induced by TIPN while providing evidence that could help unlock a better understanding of its actions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary invasive carcinoma of the breast (stage I, II, or III)
* Completed active chemotherapeutic with taxane therapy (taxotere, Taxol, Abraxane) within the last 24 months
* Established diagnosis of motor and sensory neuropathy greater or equal to 2 according to the CTCAE v 4.03 scale in spite of previous treatment with Neurontin, Cymbalta and/or Lyrica
* Read, understand, and speak English

Exclusion Criteria:

* Currently undergoing active treatment with chemotherapy (not including TKI's or other targeted therapy)
* Any acupuncture treatment for any indication within the 30 days of enrollment
* Cardiac Pacemaker
* Deformities that interfere with accurate acupuncture point locations
* Local infection at or near the acupuncture site
* Pregnant or currently lactating
* Medical History of chronic alcohol use
* Mental incapacitation or significant emotional or psychological disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-05; Primary Completion 2017-11 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in taxane induced peripheral neuropathy symptoms measured by the Patients' Global Impression of Change (PGIC) scale. | 12 Weeks
  All 18 participants will complete the PGIC scale at 6 weeks and 12 weeks. This scale will ask questions about the participants' change in activity limitations, symptoms, emotions, and overall quality of life related to their peripheral neuropathy since the beginning of treatment.
Evaluate the mechanism of acupuncture as a treatment of TIPN through quantification of inflammatory biomarkers and circulation levels of mitochondrial DNA (mtDNA) | 12 Weeks
  Approximately 8ml of blood will be collected from each participant at baseline, 6 weeks, and 12 weeks. The samples will be collected in purple top BD vacutainers.

SECONDARY OUTCOMES:
Change in quality of life using the FACT/GOG-NTX questionnaire | 12 Weeks
  Participants will complete the FACT/GOG-NTX questionnaire at baseline, 6 weeks, and 12 weeks. The questionnaire includes questions about the participants' physical, social/family, emotional, and functional well-being.
Evaluate if neuropathic mechanisms are contributing to pain measured by the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) Pain Scale | 12 Weeks
  Participants will complete the LANSS Pain Scale at baseline, 6 weeks, and 12 weeks. This pain scale involves a pain questionnaire and sensory testing to determine to determine if neuropathic mechanisms are still contributing to the participant's pain.
Change in taxane induced peripheral neuropathy related pain measured by the Brief Pain Inventory (BPI). | 12 Weeks
  Participants will complete the BPI at baseline, 6 week, and 12 week. The BPI will ask questions to detail how the pain interferes with the participants' general activity, mood, walking ability, relationships, sleep, and enjoyment of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A O'Rourke, MD, Principal Investigator — Prisma Health-Upstate; Renee J LeClair, PhD, Principal Investigator — University of South Carolina School of Medicine, Greenville
Locations (1):
- Greenville Health System Cancer Institute Center for Integrative Oncology and Survivorship, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phillips KD, Skelton WD, Hand GA. Effect of acupuncture administered in a group setting on pain and subjective peripheral neuropathy in persons with human immunodeficiency virus disease. J Altern Complement Med. 2004 Jun;10(3):449-55. doi: 10.1089/1075553041323678. PMID 15253848
- [Background] Abuaisha BB, Costanzi JB, Boulton AJ. Acupuncture for the treatment of chronic painful peripheral diabetic neuropathy: a long-term study. Diabetes Res Clin Pract. 1998 Feb;39(2):115-21. doi: 10.1016/s0168-8227(97)00123-x. PMID 9597381
- [Background] Zhang C, Ma YX, Yan Y. Clinical effects of acupuncture for diabetic peripheral neuropathy. J Tradit Chin Med. 2010 Mar;30(1):13-4. doi: 10.1016/s0254-6272(10)60003-9. PMID 20397454
- [Background] Franconi G, Manni L, Schroder S, Marchetti P, Robinson N. A systematic review of experimental and clinical acupuncture in chemotherapy-induced peripheral neuropathy. Evid Based Complement Alternat Med. 2013;2013:516916. doi: 10.1155/2013/516916. Epub 2013 Jul 24. PMID 23983788
- [Background] Carbonaro M, Escuin D, O'Brate A, Thadani-Mulero M, Giannakakou P. Microtubules regulate hypoxia-inducible factor-1alpha protein trafficking and activity: implications for taxane therapy. J Biol Chem. 2012 Apr 6;287(15):11859-69. doi: 10.1074/jbc.M112.345587. Epub 2012 Feb 24. PMID 22367210
- [Background] Hidaka M, Koga T, Kiyota H, Horiguchi T, Shi QW, Hirose K, Uchida T. Relationship between the structures of taxane derivatives and their microtubule polymerization activity. Biosci Biotechnol Biochem. 2012;76(2):349-52. doi: 10.1271/bbb.110797. Epub 2012 Feb 7. PMID 22313785
- [Background] Hu JH, Chen T, Zhuang ZH, Kong L, Yu MC, Liu Y, Zang JW, Ge BX. Feedback control of MKP-1 expression by p38. Cell Signal. 2007 Feb;19(2):393-400. doi: 10.1016/j.cellsig.2006.07.010. Epub 2006 Jul 25. PMID 16978838
- [Background] Clark IA. The advent of the cytokine storm. Immunol Cell Biol. 2007 Jun;85(4):271-3. doi: 10.1038/sj.icb.7100062. No abstract available. PMID 17551531
- [Background] Clark IA. How TNF was recognized as a key mechanism of disease. Cytokine Growth Factor Rev. 2007 Jun-Aug;18(3-4):335-43. doi: 10.1016/j.cytogfr.2007.04.002. Epub 2007 May 9. PMID 17493863
- [Background] Clark IA, Alleva LM, Budd AC, Cowden WB. Understanding the role of inflammatory cytokines in malaria and related diseases. Travel Med Infect Dis. 2008 Jan-Mar;6(1-2):67-81. doi: 10.1016/j.tmaid.2007.07.002. Epub 2007 Aug 27. PMID 18342278
- [Background] Milligan ED, Sloane EM, Langer SJ, Cruz PE, Chacur M, Spataro L, Wieseler-Frank J, Hammack SE, Maier SF, Flotte TR, Forsayeth JR, Leinwand LA, Chavez R, Watkins LR. Controlling neuropathic pain by adeno-associated virus driven production of the anti-inflammatory cytokine, interleukin-10. Mol Pain. 2005 Feb 25;1:9. doi: 10.1186/1744-8069-1-9. PMID 15813997
- [Background] Flatters SJL, Bennett GJ. Studies of peripheral sensory nerves in paclitaxel-induced painful peripheral neuropathy: evidence for mitochondrial dysfunction. Pain. 2006 Jun;122(3):245-257. doi: 10.1016/j.pain.2006.01.037. Epub 2006 Mar 13. PMID 16530964
- [Background] Kidd JF, Pilkington MF, Schell MJ, Fogarty KE, Skepper JN, Taylor CW, Thorn P. Paclitaxel affects cytosolic calcium signals by opening the mitochondrial permeability transition pore. J Biol Chem. 2002 Feb 22;277(8):6504-10. doi: 10.1074/jbc.M106802200. Epub 2001 Nov 27. PMID 11724773
- [Background] Zhang C, Jiang M, Lu A. A traditional Chinese medicine versus Western combination therapy in the treatment of rheumatoid arthritis: two-stage study protocol for a randomized controlled trial. Trials. 2011 Jun 4;12:137. doi: 10.1186/1745-6215-12-137. PMID 21639923
- [Background] Bao T, Goloubeva O, Pelser C, Porter N, Primrose J, Hester L, Sadowska M, Lapidus R, Medeiros M, Lao L, Dorsey SG, Badros AZ. A pilot study of acupuncture in treating bortezomib-induced peripheral neuropathy in patients with multiple myeloma. Integr Cancer Ther. 2014 Sep;13(5):396-404. doi: 10.1177/1534735414534729. Epub 2014 May 26. PMID 24867959
- [Background] Bennett M. The LANSS Pain Scale: the Leeds assessment of neuropathic symptoms and signs. Pain. 2001 May;92(1-2):147-57. doi: 10.1016/s0304-3959(00)00482-6. PMID 11323136
- [Background] Schoeniger-Skinner DK, Ledeboer A, Frank MG, Milligan ED, Poole S, Martin D, Maier SF, Watkins LR. Interleukin-6 mediates low-threshold mechanical allodynia induced by intrathecal HIV-1 envelope glycoprotein gp120. Brain Behav Immun. 2007 Jul;21(5):660-7. doi: 10.1016/j.bbi.2006.10.010. Epub 2007 Jan 3. PMID 17204394
- [Background] McGill MR, Sharpe MR, Williams CD, Taha M, Curry SC, Jaeschke H. The mechanism underlying acetaminophen-induced hepatotoxicity in humans and mice involves mitochondrial damage and nuclear DNA fragmentation. J Clin Invest. 2012 Apr;122(4):1574-83. doi: 10.1172/JCI59755. Epub 2012 Mar 1. PMID 22378043